CLINICAL TRIAL: NCT03128593
Title: A Phase I/II Study of JR-141 in Patients With Mucopolysaccharidosis Type II
Brief Title: A Study of JR-141 in Patients With Mucopolysaccharidosis Type II
Status: Completed | Phase: Phase 1 / Phase 2 | Type: Interventional
Sponsor: JCR Pharmaceuticals Co., Ltd. (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Sequential | Masking: None | Purpose: Treatment
Other Study IDs: JR-141-101
Record Dates: First submitted 2017-04-10; First posted 2017-04-25 (Actual); Last update posted 2022-11-14 (Actual); Status verified 2022-11

CONDITIONS: Mucopolysaccharidosis II
MeSH Terms: conditions — Mucopolysaccharidosis II

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Experimental: JR-141 (Experimental)
  Interventions: Drug: JR-141

INTERVENTIONS:
Drug: JR-141 — IV infusion (lyophilized powder), 0.01-2.0 mg/kg/week

SUMMARY:
The purpose of this study in patients with mucopolysaccharidosis type II (MPS II) is below,

* to collect the safety information of JR-141
* to evaluate the plasma pharmacokinetics of JR-141
* to explore the efficacy of JR-141 on MPS II-related central nervous system symptoms and general symptoms

ELIGIBILITY:
Inclusion Criteria:

* Patients aged 6 years or older at the time of informed consent.
* Patients diagnosed with MPS II.
* Patients who have received idursulfase (0.5 mg/kg/week) continuously for at least 12 weeks until the initial dose of JR-141.

Exclusion Criteria:

* Patients with a history of hematopoietic stem cell transplantation, excluding those who need enzyme replacement therapy even after hematopoietic stem cell transplantation.
* Patients in whom lumbar puncture cannot be performed.
* Patients who have developed serious drug allergy or hypersensitivity that is inappropriate for participation in the study.
* Patients who have received other investigational products within 4 months before enrollment in the study.

Min Age: 6 Years | Sex: Male | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 14 (Actual)
Dates: Start 2017-03-30 (Actual); Primary Completion 2017-10-04 (Actual); Study Completion 2017-10-04 (Actual)

PRIMARY OUTCOMES:
Number of participants with Adverse Events | 4 weeks
  * Adverse events
  * Laboratory tests
  * Vital signs
  * 12-lead electrocardiogram
  * Antibody
  * Infusion associated reaction

SECONDARY OUTCOMES:
Plasma Pharmacokinetic parameter [Maximum Plasma Concentration [Cmax]] | 4 weeks
  Plasma concentration of JR-141
Plasma Pharmacokinetic parameter [Area Under the Curve [AUC]] | 4 weeks
  Plasma concentration of JR-141
Urinary and serum heparan sulfate (HS) /dermatan sulfate (DS) | 4 weeks
HS/DS in CSF | 4 weeks
  JR-141 concentration in CSF
Urinary total GAG | 4 weeks
Liver and spleen volumes | 4 weeks
Cardiac function | 4 weeks

CONTACTS AND LOCATIONS:
Locations (8):
- Japan (8):
  - Gifu Clinical site, Gifu
  - Fukuoka Clinical site, Kurume
  - Tokyo clinical site1, Minato
  - Osaka Clinical site1, Osaka
  - Saitama Clinical site, Saitama
  - Tokyo clinical site2, Setagaya City
  - Osaka Clinical site2, Suita
  - Tottori Clinical site, Yonago

REFERENCES:
- [Derived] Okuyama T, Eto Y, Sakai N, Minami K, Yamamoto T, Sonoda H, Yamaoka M, Tachibana K, Hirato T, Sato Y. Iduronate-2-Sulfatase with Anti-human Transferrin Receptor Antibody for Neuropathic Mucopolysaccharidosis II: A Phase 1/2 Trial. Mol Ther. 2019 Feb 6;27(2):456-464. doi: 10.1016/j.ymthe.2018.12.005. Epub 2018 Dec 8. PMID 30595526
- See also: Iduronate-2-Sulfatase with Anti-human Transferrin Receptor Antibody for Neuropathic Mucopolysaccharidosis II: A Phase 1/2 Trial — https://pubmed.ncbi.nlm.nih.gov/30595526/